CLINICAL TRIAL: NCT00006095
Title: A Trial of Irinotecan (NSC# 616348) Plus Vincristine in Children With Solid Tumors
Brief Title: Combination Chemotherapy in Treating Children With Solid Tumors That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9971; COG-P9971 (Other: Children's Oncology Group); CCG-P9971 (Other: Children's Cancer Group); POG-9971 (Other: Pediatric Oncology Group); CDR0000068102 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-08-03; First posted 2003-05-22 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vincristine Sulfate 1.5 mg/m2/wk and Irinotecan (Experimental)
  Interventions: Drug: irinotecan hydrochloride; Drug: vincristine sulfate
- Vincristine sulfate 2.0 mg/m2/wk and Irinotecan (Experimental)
  Interventions: Drug: irinotecan hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Drug: irinotecan hydrochloride
  Other Names: CPT-11; NSC #616348
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #067574

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vincristine plus irinotecan in treating children who have solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose limiting toxicity of vincristine when administered in combination with irinotecan in children with refractory solid tumors.
* Determine the safe and tolerable phase II dose of this combination regimen in this patient population.
* Determine the pharmacokinetics of this combination regimen in these patients.
* Determine the incidence and severity of other toxicities of this combination regimen in these patients.
* Determine preliminary evidence of antitumor activity of this combination regimen in this patient population.

OUTLINE: This is a dose-escalation study of vincristine.

Patients receive vincristine IV on day 2 of the first course (day 1 of subsequent courses) and days 8, 15, 22, and 29, and irinotecan IV over 1 hour on days 1-5 and 22-26. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease receive additional courses of therapy for a maximum of 1 year.

Cohorts of 3-6 patients receive escalating doses of vincristine until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-12 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed initial diagnosis of malignant solid tumor refractory to conventional therapy or for which no effective therapy exists

  * Brain tumors allowed if not on anticonvulsants
  * Brainstem gliomas allowed without histologic diagnosis
  * Solid lymphomas allowed
* No bone marrow involvement

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* Karnofsky 50-100% if over 10 years of age
* Lansky 50-100% if 10 years of age and under

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL (transfusion allowed)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT less than 5 times normal
* Albumin at least 2 g/dL

Renal:

* Creatinine normal for age OR
* Glomerular filtration rate normal for age

Other:

* No uncontrolled infection
* No other significant systemic illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior biologic therapy and recovered
* At least 1 week since prior growth factors
* No prior stem cell transplantation

Chemotherapy:

* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No more than 2 prior chemotherapy regimens
* No other concurrent cancer chemotherapy

Endocrine therapy:

* Concurrent dexamethasone allowed in patients with CNS tumors provided dose is stable or decreasing for at least 2 weeks prior to study

Radiotherapy:

* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* No prior substantial bone marrow radiotherapy
* No prior central axis radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent anticonvulsants
* No other concurrent anticancer therapy or investigational agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2000-07; Primary Completion 2005-01 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Length of study

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S. Kretschmar, MD, Study Chair — Floating Hospital for Children at Tufts - New England Medical Center
Locations (22):
- United States (21):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia